CLINICAL TRIAL: NCT06714383
Title: A Prospective Randomized Phase Ⅱ Study of Trilaciclib Combing Chemotherapy in the Neoadjuvant Treatment of Osteosarcoma
Brief Title: Trilaciclib Combing Chemotherapy in the Neoadjuvant Treatment of Osteosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Tang Xiaodong, Dr., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMA-OS-001
Record Dates: First submitted 2024-11-23; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — trilaciclib; pirarubicin; lobaplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trilaciclib Arm (Experimental): Neoadjuvant therapy of adding Trilaciclib to Pirarubicin and Lobaplatin
  Interventions: Drug: Trilaciclib; Drug: Pirarubicin; Drug: Lobaplatin
- Control Arm (Sham Comparator): Neoadjuvant therapy of Pirarubicin and Lobaplatin
  Interventions: Drug: Pirarubicin; Drug: Lobaplatin

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib: 240mg/m2, IV, within 4 hours before each chemotherapy agent infused.
  Other Names: Cosela
  Arms: Trilaciclib Arm
Drug: Pirarubicin — Pirarubicin: 60 mg/m2，IV，d1-2
Drug: Lobaplatin — LobaplLatin: 40 mg/m2,，IV，d1

SUMMARY:
To evaluate the clinical application value in bone marrow protection of Trilaciclib in the neoadjuvant treatment of stage II/III classic osteosarcoma in combination with pirarubicin and lobaplatin.

DETAILED DESCRIPTION:
Classic osteosarcoma is the most common primary bone malignancy. At present, osteosarcoma is usually treated with preoperative chemotherapy, surgical operation and postoperative chemotherapy. Treatment with preoperative chemotherapy is also known as neoadjuvant chemotherapy. Neoadjuvant chemotherapy has brought benefits to patients, but safety concerns are inevitable. Myelosuppression is a major factor affecting the compliance of patients treated by chemotherapy. Patients with chemotherapy-induced myelosuppression(CIM) have higher rates of infection, sepsis, bleeding, and fatigue, resulting in hospitalization, hematopoietic growth factor support, blood transfusions (red blood cells and/or platelets) and even death. In addition, CIM often leads to dose reduction and delayed administration, which limits the therapeutic dose intensity and therefore affects the anti-tumor efficacy of chemotherapy.

Currently, there are no approved treatments in osteosarcoma to prevent chemotherapy-induced cell damage. Although some treatments may help to address CIM when it occurs such as blood transfusions and growth factors, these treatments are pedigree specific, being used after hematopoietic stem progenitor cells damage and could bring additional toxicity.

Trilaciclib is a highly effective, selective and temporarily reversible inhibitor of CDK4/6. The proliferation of bone marrow hematopoietic stem cells depends on CDK4/6 activity. Bone marrow hematopoietic stem cells are blocked in the G1 phase of the cell cycle after exposure to Trilaciclib before chemotherapy is given.

Therefore, this study is conducted to evaluate the clinical application value in bone marrow protection of Trilaciclib in the neoadjuvant treatment of stage II/III classic osteosarcoma in combination with pirarubicin and lobaplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed;
2. Classic osteosarcoma confirmed by histopathology (high grade);
3. Newly diagnosed stage Ⅱ-Ⅲ based on Enneking staging criteria;
4. Planned to receive neoadjuvant chemotherapy;
5. Measurable disease on CT by RECIST 1.1.
6. No antitumor system therapy received;
7. ECOG 0-1
8. Adequate organ function.
9. Females of childbearing potential as well as males and their partners must agree to use an effective form of contraception during the study and for 6 months following the last dose of study medication.

Exclusion Criteria:

1. History of malignancies of other type;
2. Allergic to study agent;
3. History of psychotropic substance abuse, alcohol or drug use;
4. The researchers considered inappropriate to join the study of any cause.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3/4 neutropenia | up to 30 days
  Incidence of grade 3/4 neutropenia up to 30 days

SECONDARY OUTCOMES:
Duration of grade 3/4 neutropenia | up to 30 days
  Duration of grade 3/4 neutropenia up to 30 days
Incidence of grade 3/4 thrombocytopenia | up to 30 days
  Incidence of grade 3/4 thrombocytopenia up to 30 days
Incidence of grade 3 or 4 anemia | up to 30 days
  Incidence of grade 3 or 4 anemia up to 30 days
Incidence of febrile neutropenia | up to 30 days
  Incidence of febrile neutropenia up to 30 days
Usage of granulocyte colony-stimulating factor (G-CSF) | up to 30 days
  Utilization rate of granulocyte colony-stimulating factor (G-CSF) up to 30 days
Usage of Thrombopoietin (TPO) | up to 30 days
  Utilization rate of Thrombopoietin (TPO) up to 30 days
Usage of Erythropoietin (ESA) | up to 30 days
  Utilization rate of Erythropoietin (ESA) up to 30 days
Incidence of platelet transfusion | up to 30 days
  Incidence of platelet transfusion up to 30 days
Incidence of red blood cell transfusion | up to 30 days
  Incidence of red blood cell transfusion up to 30 days
Usage of ferralia | up to 30 days
  Utilization rate of ferralia up to 30 days
chemotherapy dose reduction of any cause | up to 30 days
  chemotherapy dose reduction rate of any cause up to 30 days
AE adverse event adverse event adverse event | up to 30 days
  adverse event
SAE | up to 30 days
  serious adverse event serious adverse event serious adverse event Serious Adverse Event
Termination of treatment caused by AE/SAE | up to 30 days
  Termination of treatment rate caused by AE/SAE

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China